CLINICAL TRIAL: NCT01649011
Title: Validation of a Translation Into Spanish of the Oswestry Disability Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Galvan Ernesto Eduardo, Galvan Ernesto Eduardo MD, MSc, Principal investigator, American British Cowdray Medical Center
Other Study IDs: ABC-ODI-12-2012
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Low Back Pain
Keywords: Oswestry Disability Index; ODI; Roland Morris Disability Questionnaire; RMDQ
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Scores of the ODI and RMQ for low back pain
  Interventions: Behavioral: Application of the initial evaluation; Behavioral: Final application of scales

INTERVENTIONS:
Behavioral: Application of the initial evaluation — Initial evaluation involves the application of the previously spanish validated Rolland Morris Questionnaire and the new spanish Oswestry Disability Index
Behavioral: Final application of scales — Application of the previously spanish validated version of the RMQ and the new spanish translation of the ODI 2 weeks after initial evaluation

SUMMARY:
The purpose of the study is to validate in Mexico a spanish translation of the 2.1a Oswestry Disability Index (ODI) version in patients with low back pain.

Internal consistency, reproducibility and reliability will be addressed scoring the results of the translated version at two time frames. A previously spanish validated translation of the of the Roland Morris Disability Questionnaire (RMDQ) will be used to compare and evaluate both versions.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most frequent ailments in industrialized countries, with a lifetime prevalence of more than 70%, and is responsible for a major portion of work absenteeism. Measuring disability is important in LBP. First, as an outcome measure, it is an important indicator of the quality of life of the patient. The Oswestry Disability Index (ODI) and the Roland Morris Disability Questionnaire (RMDQ) have emerged as the most commonly recommended condition specific outcome measures for spinal disorders.

The development of the ODI was initiated by John O'Brien in 1976. The index was designed as a measure for both assessment and outcome on patients with low back pain. The questionnaire can be completed in less than 5 minutes and scored in less than 1 minute. Version 1.0 of the questionnaire was published in 1980 and widely disseminated after the 1981 meeting of the International Society for The Study of the Lumbar Spine (ISSLS) in Paris. A new ODI version was adapted in 1989 by the Chiropractic College in England. The American Academy of Orthopedic Surgeons and other spine associations adapted the ODI 1.0 version in 1996 omitting categories 1, 8 and 9. This version is included in the assessment protocol proposed by the Musculoskeletal Outcomes Data Evaluation and Management System (MODEMS), which brings together the main international spine associations. Version 2.0 was modified by the Medical Research Council Group in the UK in 1996 (16) and they omitted the word "painkillers" in the first category. Version 2.1a is the most recent and recommended by its author. In this version a section called previous treatment appears, which is not taken into account for scoring. The score can be obtained for its clinical use after permission at: http://www.mapi-trust.org/.

The RMDQ is a health status measure designed to be completed by patients to assess physical disability due to low back pain. It was designed for use in research (e.g., as an outcome measure for clinical trials) but has also been found useful for monitoring patients in clinical practice. Was derived from the Sickness Impact Profile (SIP), which is a 136 item health status measure covering all aspects of physical and mental function. Twenty four items were selected from the SIP by the original authors. It is simple, fast, and can be filled out by the patient. The patient must mark each item that applies to his or her current LBP. Scoring is also simple and fast; each checked item receives a score of 1, so scores range between 0 (no disability caused by LBP) and 24 (the maximum possible disability). To date only one version has been translated to Spanish and was published in 2002 by Kovacks FM, et al.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or chronic low back pain
* With or without previous back surgery

Exclusion Criteria:

* Visual or mentally impaired

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Low back pain scored by the translated and proposed version of the ODI | Initial evaluation and 2 weeks after
  The objective of this outcome measure is to evaluate the ability of the translated ODI version to measure changes in time on patients with low back pain. The score will be registered 2 times with 3 weeks apart

SECONDARY OUTCOMES:
Low back pain scored by the RMQ spanish version | Initial evaluation and 2 weeks after
  The RMQ will be administered at the same time that the proposed translated ODI version, at the beginning of the study and 3 weeks later. The RMQ was previously translated and validated to spanish, and will work like a reference to evaluate the reproducibility of any change in the score obtained by the ODI spanish version.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto E Galvan Hernandez, MD, MSc, Principal Investigator — American British Cowdray Medical Center
Locations (1):
- American British Cowdray Medical Center, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Kovacs FM, Llobera J, Gil Del Real MT, Abraira V, Gestoso M, Fernandez C, Primaria Group KA. Validation of the spanish version of the Roland-Morris questionnaire. Spine (Phila Pa 1976). 2002 Mar 1;27(5):538-42. doi: 10.1097/00007632-200203010-00016. PMID 11880841
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727